CLINICAL TRIAL: NCT05559554
Title: A Phase I Study to Evaluate the Similarity of Pharmacokinetic (PK) in AK104 (a PD-1/CTLA-4 Bispecific Antibody) With Different Manufacturing Process in Healthy Chinese Male Subjects
Brief Title: A Study to Evaluate the PK Similarity of AK104 in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AK104-102
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy Male Subjects
Keywords: AK104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 (after the change) (Experimental): Drug: AK104 (after the change) Dose 1 and dose 2, will be administrated intravenously in 60±10 minutes.
  Interventions: Drug: AK104 (after the change)
- AK104 (before the change) (Active Comparator): Drug: AK104 (before the change) Dose 1 and dose 2, will be administrated intravenously in 60±10 minutes.
  Interventions: Drug: AK104 (before the change)

INTERVENTIONS:
Drug: AK104 (before the change) — Dose 1 and dose 2 in pilot study, and recommended dose in pivotal study.
  Arms: AK104 (before the change)
Drug: AK104 (after the change) — Dose 1 and dose 2 in pilot study, and recommended dose in pivotal study.
  Arms: AK104 (after the change)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic similarity of AK104 with different manufacturing process in healthy male subjects. Another purpose is to determine safety, and immunogenicity of AK104 with different manufacturing process.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 to 45;
2. Body Mass Index (BMI) is 19.0~28.0 kg/m2, and body weight is 50.0~80.0kg ;
3. Signing informed consent form before the trial and having a full understanding of the trial content, process and possible adverse reactions;
4. Able to complete the study according to the requirements of the study protocol.

Exclusion Criteria:

1. Those with a history of digestive tract, respiratory, cardiovascular, endocrine, urinary, neurological, hematological, metabolic and other systemic diseases;
2. Those with a history of autoimmune diseases;
3. Those with a history of malignant tumor, unless it is a skin squamous cell carcinoma, basal cell carcinoma or cervical cancer in situ that has been successfully resected and has no evidence of metastasis;
4. Regular drinkers within 6 months prior to screening;
5. Those who are suspected or confirmed to be allergic or have had severe drug or food allergy reactions in the past, have a clear history of allergies and/or are allergic to the study drug or its components after inquiries;
6. Those who have used anti-PD-1/PD-L1 or/and anti-CTLA-4 drugs in the past;
7. Those who have been vaccinated with live or attenuated-live vaccines within 3 months before screening, or who are expected to receive vaccines during the study period;
8. Those who lost blood, donated blood or received any blood product transfusion of ≥400 ml within 3 months before screening;
9. Those who received major surgery or hospitalization due to illness within 3 months before screening;
10. Abnormal laboratory tests with clinical significance at screening;
11. Positive drug screening result;
12. Have a childbirth plan within 6 months from the screening period to the trial drug administration, or who are unwilling to take the contraceptive measures specified in the protocol during the trial period.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Pilot study: Adverse Events (AEs) | Up to day 30
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Pivotal study: Area under the plasma concentration-time curve (AUC0-infinity) | From pre-dose to day 29

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t) | From pre-dose to day 29
Maximum plasma concentration (Cmax) | From pre-dose to day 29
Volume of distribution (Vd) | From pre-dose to day 29
Clearance (CL) | From pre-dose to day 29
Ratio of AUC0-t/AUC0-infinity | From pre-dose to day 29
Time to maximum concentration (Tmax) | From pre-dose to day 29
Half-life (t1/2) | From pre-dose to day 29
Anti-drug Antibody (ADA) | From pre-dose to day 29
  Number and percentage of subjects with detectable ADA

CONTACTS AND LOCATIONS:
Overall Officials: Xin Li, MD, Principal Investigator — The Third Hospital of Changsha
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China